CLINICAL TRIAL: NCT05423288
Title: Textbook Outcome in Distal Pancreatectomy: a Multicenter Study
Brief Title: Textbook Outcome in Distal Pancreatectomy
Acronym: TO-ERPANDIS
Status: Completed | Type: Observational
Sponsor: Universidad de Extremadura (Other)
Responsible Party: Principal Investigator, Gerardo Blanco-Fernández, Professor, Universidad de Extremadura
Other Study IDs: UE-CHUB-002-2022
Record Dates: First submitted 2022-06-13; First posted 2022-06-21 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Distal Pancreatectomy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Distal pancreatectomy (DP) — Any scheduled distal pancreatectomy performed for any diagnosis

SUMMARY:
The auditing of results and improving the quality of care are key aspects of surgical activity. Patients, hospitals and health institutions need information on the results obtained with specific procedures. The most commonly used method to assess quality of care is the measurement of postoperative complications, hospital stay, and readmission rates. Other assessment tools such as benchmarking allow comparisons to be made between centers.

In 2013, Kolfschoten et al. introduced a new measure called textbook outcome (TO), a single indicator that combines several traditional care measures: the absence of postoperative complications, no prolongation of hospital stay (< 75th percentile), no mortality and no readmissions. All these parameters must be fulfilled in order to achieve textbook outcome (TO).

The investigators analyze the achievement of TO in a multicenter DP database using a specific TO for distal pancreatectomy (DP) (TO-DP) which includes clinically-relevant pancreatic fistula (grade B/C).

DETAILED DESCRIPTION:
Retrospective, multicenter, observational study of prospectively recorded data regarding DP carried out at 8 hepato-pancreato-biliary (HPB) surgical units between 1 January 2008 and 31 December 2018. Five are high-volume HPB units at level 3 hospitals in Spain, the highest level in our country; one is the reference center for HPB surgery and transplantation in Puerto Rico, and two are level 2 hospitals in Spain. Six authors are UEMS HPB Board Certificate.

Each participating center appointed a local manager to carry out the data collection and to liaise with the overall study coordinator. All the data were collected by the local managers at each hospital, and the project coordinator had access to medical data only.

The study has been conducted in accordance with the Declaration of Helsinki (2013), and was approved by the institutional ethics committee of the Hospital Universitario de Guadalajara (CEIm: 2018.17.EO) (27-11-2018). The need to obtain patients' informed consent was waived since the study was retrospective and observational, and entailed no risk.

Inclusion criteria were any scheduled PD performed for any diagnosis and age >18 years. Exclusion criteria were PD with celiac trunk resection. The suspected preoperative diagnosis was based on CT, MRI and EUS plus biopsy. The surgical approach was either open or laparoscopic, with or without spleen preservation. Complications were assessed at 90 days using the Clavien-Dindo (CD) classification, and those defined as Clavien-Dindo grade III or IV were considered major; they were recorded from the electronic medical and nursing notes or clinical histories of each patient. For complications specific to pancreatic surgery, the definitions of the International Study Group on Pancreatic Surgery (ISGPS) for delayed gastric emptying, post-pancreatic hemorrhage and pancreatic fistula were used. The resection margins of the specimen were categorized according to the Royal College of Pathologists definitions: R0 (margin to the tumor ≥ 1mm), R1 (margin to the tumor < 1mm) and R2 (macroscopically positive margin). Invasive tumors were staged according to the TNM classification (8th ed.). The follow-up scheme applied at all centers comprised 3 or 6-month outpatient clinic visits during the first five years depending on diagnosis, including tumor marker assessment and CT/MRI, and after five years an annual visit (in non-invasive cases). TO-DP was defined including classical variables: hospital stay p < 75, Clavien-Dindo complication Grade ≥ 3, in-hospital mortality and re-admission within 90 days, and pancreatic fistula (grade B or C).

Variables

The following variables were included in the study. Epidemiological variables: age, sex, past abdominal surgeries, medication and ASA; Clinical variables: symptoms, serological tests, leukocytes, hemoglobin (gr/dl); Radiological/diagnostic variables: vascular infiltration (arterial and venous) and preoperative biopsy; Surgical variables: type of approach (open/laparoscopy), spleen preservation, associated organ resection, intraoperative red blood cell (p-RBC) transfusion; Postoperative course: morbidity and mortality (according to the CD classification), pancreatic fistula, postoperative hemorrhage and delayed gastric emptying (if present, classified according to the ISGPS classification), hospital stay and readmissions. The histological data recorded were tumor size and size of resected pancreas.

Statistical analysis

Descriptive statistics were calculated using frequencies and percentages for categorical data, and medians and interquartile ranges (IQR) for continuous data. Differences between groups in the case of quantitative variables were analyzed using the non-parametric Mann-Whitney U test, and differences between percentages or frequencies using Pearson's Chi-square test. A p value < 0.05 was considered statistically significant. Logistical regression analyses were performed to investigate possible relationships between the characteristics of the variables and the achievement of TO. First, univariate analysis was used to explore the unadjusted association between each variable and outcome. Then, variables with a p value < 0.10 were included in the multivariate analysis. Calculations were performed using the programs Microsoft Excel for Mac, version 16.49 and SPSS for Mac, version 26.0 (SPSS Inc., Chicago, Illinois, USA).

ELIGIBILITY:
Inclusion Criteria:

* Any distal pancreatectomía performed for any diagnosis

Exclusion Criteria:

* Distal pancreatectomy with celiac trunk resection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients operated on distal pancreatectomy. The surgical approach was either open or laparoscopic, with or without spleen preservation
Sampling Method: Non-Probability Sample
Enrollment: 450 (Actual)
Dates: Start 2008-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Mortality | 90 days
  No postoperative mortality within 90 days after surgical procedure
Morbidity | 90 days
  No major complications within 90 days after surgical procedure
Re-admission | 90 days
  No re-admissions within 90 days after surgical procedure

CONTACTS AND LOCATIONS:
Overall Officials: Gerardo Blanco-Fernández, MD, PhD, Principal Investigator — Universidad de Extremadura

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mehta R, Tsilimigras DI, Pawlik TM. Assessment of Magnet status and Textbook Outcomes among medicare beneficiaries undergoing hepato-pancreatic surgery for cancer. J Surg Oncol. 2021 Sep;124(3):334-342. doi: 10.1002/jso.26521. Epub 2021 May 7. PMID 33961716
- [Background] Ramia JM, Soria-Aledo V. Textbook outcome: A new quality tool. Cir Esp (Engl Ed). 2021 Jul 6:S0009-739X(21)00215-3. doi: 10.1016/j.ciresp.2021.06.002. Online ahead of print. No abstract available. English, Spanish. PMID 34243935
- [Background] de la Plaza Llamas R, Ramia Angel JM, Bellon JM, Arteaga Peralta V, Garcia Amador C, Lopez Marcano AJ, Medina Velasco AA, Gonzalez Sierra B, Manuel Vazquez A. Clinical Validation of the Comprehensive Complication Index as a Measure of Postoperative Morbidity at a Surgical Department: A Prospective Study. Ann Surg. 2018 Nov;268(5):838-844. doi: 10.1097/SLA.0000000000002839. PMID 30303875
- [Background] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542